CLINICAL TRIAL: NCT03756246
Title: Influenza Vaccine as a Novel Experimental Model of the Behavioral Immune Response in Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018030078
Record Dates: First submitted 2018-11-14; First posted 2018-11-28 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Depression; Healthy
Keywords: depression; Major Depressive Disorder; depressive
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Both healthy and depressed arms will receive the influenza vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Depression Subjects: Influenza Vaccine (Experimental): Subjects will receive a quadrivalent inactivated influenza vaccine, for the appropriate season/year of enrollment. The vaccine will be administered by the PI or similarly trained clinician, into the deltoid muscle as directed
  Interventions: Biological: Influenza Vaccine
- Healthy Subjects: Influenza Vaccine (Active Comparator): Subjects will receive a quadrivalent inactivated influenza vaccine, for the appropriate season/year of enrollment. The vaccine will be administered by the PI or similarly trained clinician, into the deltoid muscle as directed
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — The appropriate quadrivalent influenza vaccine for the give year will be given to subjects.
  Other Names: flu shot; flu vaccine

SUMMARY:
The purpose of this study is to determine differences between the immune responses in healthy and depressed people. Participants will receive the influenza vaccine and their responses will be monitored. This study will recruit 15 healthy and 60 depressed participants.

DETAILED DESCRIPTION:
The purpose of this study is to determine differences between the immune responses in healthy and depressed people. Specifically subjects are provided a mild immune stimulus, an influenza vaccine, and their responses are monitored. The goals are to determine whether patients with depression experience a temporary worsening of mood in response to the stimulus and whether this is associated with measurable differences in the cytokine response to the vaccine. Additionally, patients with depression may be less likely to mount a successful antibody response to vaccination as healthy people based on circumstantial evidence, and this study will assess whether this the case.

This study aims to recruit a sample of 15 healthy and 60 depressed participants. The 15 healthy participants will be age and gender matched to the first 15 depressed participants recruited. Three more sets of age and gender matched depressed subjects will be recruited. This will result in 15 sets of "quintuplets" (4 depressed and one healthy), that are matched by age and gender. The study consists of four visits. The first visit is the baseline assessment where participants will receive the influenza vaccine. Participants will then return 1, 3 and 28 days after receiving the vaccine to assess their responses.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all subjects

* Adults age 18-60
* Able to provide written informed consent directly, without use of a proxy
* Able to speak and write in English sufficiently to undergo consent and to complete self reports

Inclusion Criteria for depressed subjects

* Currently meets criteria for a Depressive Episode and a diagnosis of MDD according Mini International Neuropsychiatric Interview (MINI)
* Depressive severity of ≥ 12 on the Quick Inventory of Depression Symptomatology, Clinician Rated (QIDS-C), corresponding to more than mild depression severity, but <21, indicating not severe

Inclusion Criteria for healthy Subjects

* No lifetime Axis I diagnosis on the MINI
* QIDS-SR score <6 indicating no depression
* CRP at screening of <1mg/L.

Exclusion Criteria:

Exclusion Criteria for all subjects

* Active, unstable, or serious medical illness (e.g. requiring urgent out-patient or higher level of care) as determined by history and lab examination at screening. For example, subjects with untreated cardiovascular disease (blood pressure above 140/80 on repeated measurements, history of cardiac event without medical follow up) or untreated diabetes (based on symptoms and elevated fasting blood sugar at screening) will be excluded.
* Taking medications that have a significant effect on the immune system. This includes daily Non-steroidal Anti-inflammatory medications (NSAIDs). As needed NSAIDs will not be exclusionary but subjects will be asked to refrain from NSAID usage for 48 hours prior to the vaccination visit and through the day 3 visit.
* Has received the influenza vaccine for the current season or within the last 12 months
* Infection with fever or otherwise clinically significant in the last two weeks. Subjects with elevated white blood cell count at screening will also be excluded.
* Current and within the last 3 months meeting criteria for tobacco use disorder.
* Previous severe adverse event associated with IIV
* History of allergy to any component of the IIV
* History of Guillain-Barre Syndrome
* Pregnancy
* Otherwise judged unable to comply with study procedures or unsafe to participate by study clinician

Exclusion Criteria for Depressed Subjects

* Life-time history of mania, hypomania, or psychosis on the MINI
* Meets or has met criteria for substance abuse or dependence in the last 6 months (3 months for nicotine)
* Meets or has met criteria for any eating disorder in the last 6 months
* Baseline suicidal ideation above "passive" defined as thoughts of death or dying (e.g. wish for natural death) without thoughts of active methods (e.g. overdose) or intent to die, as determined using the Concise Health Risk Tracking Scale (CHRT) (assessment interval "the last week") and clinician interview.

No Exclusion Criteria for Healthy Subjects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedules Score | 1 Day
  We will compute change in scores on the PANAS-x subscales between baseline and day 1. Self reported assessment that contains both positive and negative words and phrases that describe different feelings and emotions. Subjects read each item and mark the appropriate answer for how they feel right now as they fill out the form. Possible answers and the associated score are: (1) Not at all, (2) A little, (3) Moderately, (4) Quite a bit, (5) Extremely. To rate, responses to items in each scale are summed. The scales in the PANAS are listed below with the number of items in that scale in parentheses followed by the total range of the scale.
  General Dimensions Negative Affect (10) 10-50 General Dimensions of Positive Affect (10) 10-50 Negative Emotion Fear (6) 6-30 Hostility (6): 6-30 Guilt (6): 6-30 Sadness (5) 5- 25 Positive Emotion Joviality (8) 8-40 Self-Assurance (6) 6-30 Attentiveness (4) 4-20 Other Affective States Shyness (4) 4-20 Fatigue (4) 4-20 Serenity (3) 3-15

SECONDARY OUTCOMES:
Change in Cytokine Concentration (pg/mL) | 3 Days
  We will compute differences in cytokine (IFN- α, IFN-y, IL-6, IL1-β and TNF-α) values for each subject between baseline and day 1 and days 1 and 3. Using OLS regression we will compute regressions between hypothesis appropriate time points using baseline CRP, QIDS, PANAS score and BMI as covariates.
Difference in PGE4/LipoxinA4 Ratio | 3 Days
  After determining the difference in the PGE4/LipoxinA4 ratio between days 1 and 3, we will perform a similar regression.
Tryptophan Metabolites | 1 Day
  We will calculate difference between baseline and day 1 in the KYN/TRP and KYNA/QUIN ratios and us them in regression models as above, correcting for two tests.
HPA Axis | 3 Days
  To test the hypothesis that ACTH/cortisol affects peak inflammatory cytokine levels in MDD, we will use similar OLS regression models including HPA-axis response as a covariate and examining its interaction with cytokines as the dependent variables.

OTHER OUTCOMES:
Fold Change | 28 Days
  : Fold change from pre- to 28 days post-vaccine will be calculated for each of the three influenza strains targeted by the vaccine. Fold change > 4 to any one of the three strains will be considered "success." Proportion of successful vaccination will be compared between HC and MDD using a linear model adjusted for age and pre-vaccination titer, which have been shown to affect antibody response.

CONTACTS AND LOCATIONS:
Locations (1):
- Marisa Toups, Austin, Texas, United States